CLINICAL TRIAL: NCT04320043
Title: The Risk of Adjacent Segment Disease After Anterior Cervical Discectomy With Fusion for Cervical Degenerative Disc Disease
Brief Title: Adjacent Segment Disease After Anterior Cervical Decompression Surgery
Acronym: ASDafterACDF
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METCZ2020004
Record Dates: First submitted 2020-03-11; First posted 2020-03-24 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Adjacent Segment Disease; Cervical Myelopathy; Cervical Radiculopathy; Degenerative Disc Disease
Keywords: Adjacent Segment Disease; Anterior Cervical Discectomy; Anterior Cervical Discectomy with Fusion; ACD; ACDF; Cervical Radiculopathy; Cervical Myelopathy; Degenerative Disc Disease; Discectomy; Corpectomy
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anterior cervical decompression surgery: Adult patients who underwent anterior cervical decompression surgery for radiculopathy and/or myelopathy due to cervical degenerative disc disease. Patients underwent one of the following interventions: ACD, ACDF, ACDF with plating or corpectomy.
  Interventions: Procedure: Anterior cervical decompression

INTERVENTIONS:
Procedure: Anterior cervical decompression — Any of the following anterior surgical techniques used to decompress the cervical nerve roots or spinal cord; corpectomy, Anterior Cervical Discectomy (ACD), Anterior Cervical Decompression and Fusion (ACDF) or ACDF with Plating

SUMMARY:
Radiculopathy and/or myelopathy due to cervical degenerative disc disease are increasingly common pathologies in our ageing population. Both can be treated non-surgically or surgically. The most commonly used neurosurgical treatment is anterior cervical discectomy with or without fusion. The goal is to achieve neural decompression of the operated segment in both procedures. However, due to this fusion and reduced mobility of the cervical spine at the level of the intervention, adjacent segment disease may occur. This can lead to new symptoms like radiculopathy and/or myelopathy at an adjacent level which requires reoperation in about 2/3 of patients. Reoperations are burdensome for patients and have a socio-economic impact due to the costs of hospital admissions, operations, and secondary costs such as work-absenteeism. The primary objective of this retrospective study is to determine the occurrence of adjacent segment disease after a single- or multi-level anterior cervical discectomy with fusion procedure for radiculopathy and/or myelopathy in the investigators' centre and to compare this to the incidence in literature. The investigators also look at the risk of adjacent segment disease after different anterior surgical techniques, such as anterior cervical discectomy, anterior cervical discectomy with fusion and plating, and corpectomy. As a secondary outcome they aim to determine risk factors predicting the occurrence of adjacent segment disease.

DETAILED DESCRIPTION:
1. SUMMARY Radiculopathy and/or myelopathy due to cervical degenerative disc disease are increasingly common pathologies in our ageing population. Both can be treated non-surgically or surgically. The most commonly used neurosurgical treatment is anterior cervical discectomy with or without fusion. The goal is to achieve neural decompression of the operated segment in both procedures. However, due to this fusion and reduced mobility of the cervical spine at the level of the intervention, adjacent segment disease may occur. This can lead to new symptoms like radiculopathy and/or myelopathy at an adjacent level which requires reoperation in about 2/3 of patients. Reoperations are burdensome for patients and have a socio-economic impact due to the costs of hospital admissions, operations, and secondary costs such as work-absenteeism. The primary objective of this retrospective study is to determine the occurrence of adjacent segment disease after a single- or multi-level anterior cervical discectomy with fusion procedure for radiculopathy and/or myelopathy in the investigators' centre and to compare this to the incidence in literature. The investigators also look at the risk of adjacent segment disease after different anterior surgical techniques, such as anterior cervical discectomy, anterior cervical discectomy with fusion and plating, and corpectomy. As a secondary outcome they aim to determine risk factors predicting the occurrence of adjacent segment disease.
2. INTRODUCTION AND RATIONALE Radiculopathy and myelopathy are pathologies which, amongst others, occur due to cervical disc herniation or spondylosis, also known as cervical degenerative disc disease (CDDD). Radiculopathy has been estimated to affect around 100 per 100.000 males and 60 per 100.000 females in the general population. The incidence of myelopathy is estimated to be 4 per 100.000 in the general population. The consequences of CDDD can be severe and can disable patients to an extent that it impairs working ability. Therefore, it leads to a significant socio-economic burden of disease.

   Cervical radiculopathy is caused by compression of the cervical nerve roots as they exit the vertebral column through the neuroforamina. Patients present with radiating pain in the arm in the corresponding dermatome, weakness and/or sensory loss, with or without associated neck pain. Cervical myelopathy is caused by a central canal stenosis, which causes compression of the spinal cord itself. Damage to the central nervous system at this level can cause loss of coordination, motor, and sensory function of both arms and legs. Treatment for radiculopathy and/or myelopathy due to CDDD can be non-surgical or surgical. The majority of patients with radiculopathy respond well to non-surgical treatment options, such as physical therapy, a neck collar, analgesic or anti-inflammatory medication. Surgery can be considered in cases of insufficient relief with these non-surgical treatment options. The reported surgery rates range from 8% to 35%. When patients have mild myelopathy, which does not progress clinically, non-surgical treatment with frequent follow-up is an option, however, controversy exists. Others suggest surgical treatment with mild myelopathy, to prevent deterioration of symptoms. Surgery is recommended in patients with moderate and severe degenerative cervical myelopathy (DCM) or with rapid clinical deterioration.

   Both anterior and posterior surgical techniques are used to treat radiculopathy and/or myelopathy. No clear consensus exists on which anterior technique is superior. Depending on country, centre and surgeon, different approaches are used, mostly based on experience. Anterior cervical discectomy with (ACDF) or without fusion (ACD) are the most commonly used interventions for CDDD since the compression is often located on the anterior side. Alternatives are corpectomy or ACDF with plating. In the investigators' centre ACDF is the procedure of choice in most patients with single- or multilevel CDDD and radiculopathy and/or myelopathy. ACD and ACDF both have good short-term clinical results. However, in the long-term patient satisfaction drops, which is probably for a large part due to adjacent segment disease (ASD). This occurs in approximately 25% of patients during 10 years follow-up and over 2/3 of these patients need additional surgery. ASD is thought to be a consequence of fusion of two or more vertebra which eliminates mobility at the level of the intervention. Adjacent levels compensate for this reduced mobility by increasing their mobility and thus increasing their risk at disc degeneration. This risk is not only determined by the biomechanical stress on the adjacent level caused by fusion. Changes in the anatomy at the adjacent level with the initial surgery and the natural course of the adjacent disc also plays a role.

   Anterior cervical discectomy with arthroplasty (ACDA) was developed in an effort to reduce the incidence of ASD by preserving physiological motion in the operated segment. ACDA has been confirmed to ACDF for treatment of two-level CDDD, a significantly lower re-operation rate in the ACDA group compared to the ACDF group was found after two years (3.1% versus 11.4%, respectively). Re-operation rates for ACDA and ACDF after 7 years were compared. They reported reoperation rates of 3.7% for ACDA versus 13.6% for ACDF in single-level CDDD patients. The rate of reoperation was also significantly lower in the two-level ACDA group compared to ACDF, with rates of subsequent surgery at the index level of 4.4% versus 16.2% and rates of adjacent level surgery of 4.4% versus 11.3%, respectively. In a systematic review from 2017 multilevel ACDA was proven at least as safe and effective as ACDF, with preservation of cervical motion and potentially with fewer reoperations expected.

   The goal of this study is to determine the risk of ASD after ACD(F) for radiculopathy and/or myelopathy in the study population, and to compare this to the rates reported in literature. The expectation is that the occurrence in the study population is similar to the occurrence in the general population.

   The investigators will also look at the risk of ASD after different anterior surgical techniques, e.g. ACDF with plating, ACD, corpectomy. These are less commonly used procedures in the study centre. Due to the biomechanical stress induced by fusion, higher rates of ASD are expected after ACDF with plating and corpectomy than after ACDF or ACD. As a secondary outcome the investigators aim to determine risk factors predicting the occurrence of adjacent segment disease. Age and degeneration of the cervical spine are expected to play a role. Therefore, baseline characteristics will be assessed and the Kellgren's score on pre-operative X-rays will be determined.
3. METHODS 3.1 Study design A retrospective cohort study will be conducted in the Zuyderland Medical Center, Heerlen and Maastricht UMC+, Maastricht. Patients undergoing anterior cervical decompression surgery in the past 10 years will be analysed. The occurrence of ASD will be the primary outcome. Baseline characteristics will be assessed to determine predictive factors for ASD. Data will be assessed in the electronic patient files and a database will be constructed. This study is expected to take about a year from the METC approval to submitting the article.

   3.2 Study selection 3.2.1 Study population and selection The study population consists of adult patients who underwent anterior cervical decompression for radiculopathy and/or myelopathy due to CDDD in the Zuyderland MC Heerlen or MUMC+ Maastricht in the past 10 years. The following anterior surgical decompression techniques will be included; ACD, ACDF, ACDF with plating, and corpectomy. The data manager for Zuyderland Medical Center and Maastricht UMC+ will conduct a search of the electronic patients records in this period using DBC/DOT codes for above mentioned neurosurgical interventions.

   3.2.2 Sample size There will be around 100 patients per year that can be included in the study which gives an estimated total sample size of approximately 1000 patients. As this is a retrospective cohort study, the number of patients that can be included is set. With the given sample size and power, the smallest possible difference this study can show could be calculated. However, in this study this is not relevant. Based on previous studies, as shown in the hypothesis, an incidence between 10% and 20% is expected.

   With a sample size of 1000 and an incidence of 10%, the 95% confidence interval (including continuity) is 8,25%-12,07% (width 3,82%). With a sample size of 1000 and an incidence of 20%, the 95% confidence interval (including continuity) is 17,59-22,64% (width 5,05%). Concluding: with an incidence of 10-20% and a sample size of 1000, the width of the confidence intervals will be 3,82-5,05%. This can be considered small, which indicates a sufficient sample size.

   To examine the effect of parameters that may have an influence on the occurrence of ASD, 10 events and 10 non-events are needed per parameter. If the incidence were to be 10% with a sample size of 1000, there are 100 events. This means 10 parameters can be included in the analysis.

   3.3 Data selection Baseline data will be collected from the electronic patient file (EPD). Treatment data such as the indication and level of surgery will be documented, as well as complications related and not-related to the surgery.

   When interpreting the clinical outcome after the surgery, the following has to be taken into account. For radiculopathy, a good clinical outcome means improvement. A poor outcome is either stabilisation or deterioration. For myelopathy a good outcome is stabilisation (or in some cases improvement) and only deterioration is considered as a poor outcome. Baseline and treatment data will be collected to evaluate whether they attribute to the risk on developing ASD.

   Baseline data
   * Age (years)
   * Gender (male/female)
   * Body Mass Index (BMI) (kg/m2)
   * Smoking (yes/no)
   * Pre-operative duration of symptoms (weeks)
   * Indication (myelopathy/radiculopathy/both)
   * Level of CDDD (C3-C4, C4-C5, C5-C6, C6-C7, C7-Th1)
   * Post-operative use of pain medication (yes/no)
   * Kellgren's score (0-4)

   Treatment data
   * Intervention (ACDF/ACDF with plating/ACD/corpectomy)
   * Level of surgery (C3-C4, C4-C5, C5-C6, C6-C7, C7-Th1)
   * Single or multilevel (1-level/2-level/more than 2 levels)
   * Follow-up duration (months)

   Outcome parameters
   * Radiculopathy (good/poor)
   * Myelopathy (good/poor)
   * Re-operation for ASD (yes/no)
   * New symptoms (yes/no, radiculopathy/myelopathy/both, level)

   Complications
   * Related to surgery (none/failure of treatment/death)
   * Other (death)

   3.4 Data analysis Statistical analyses will be carried out using IBM SPSS statistics 25. Summary statistics will be calculated for demographic, treatment and outcome variables. T-tests will be used for continuous variables. X2 tests will be used for categorical variables. ANOVA-analyses will be used is case of more than two groups. Analyses will be two-sided. P values of < 0.05 will be considered significant differences.

   Descriptive statistics will be used to assess the incidence of ASD in the study population.

   A logistic regression analysis will be performed with regard to the outcome parameters. A survival analysis will be performed to evaluate the risk factors for ASD over time.

   3.5 Data management A coded excel file will be created with obtained patient data. The key to the code will be stored separately and safely in the MUMC+. Information and results will be stored in SPSS where only patient numbers will be mentioned. Names and other personal information, such as date of birth will be left out of this file. Data and results will be stored on password protected computers and a hard drive secured by the hospital. The files are only available for the investigators involved in the study (Dr. A. Smeets, Drs. V. Schuermans and Drs. N. Wijsen) and will not leave the hospital. Handling of personal data will comply with the Dutch Personal Data Protection Act (Wbp).

   Data will be stored for 15 years in the concerning centre.
4. ETHICAL CONSIDERATIONS The study protocol will be submitted to the Medisch Ethische Toetsings Commissie van Zuyderland en Zuyd Hogeschool Zuderland The Medical Research Involving Human Subject Act does not apply to the above-mentioned study (niet WMO-plichtig onderzoek).

   The 'geen bezwaarregeling"; is applicable seen the impossible workload of contacting an estimated 800 patients to ask for informed consent. Moreover, a large amount of these patients might have changed contact information or may have deceased. The patients and their lives will not be negatively influenced seen all data is anonymized. When patients are contacted, they are asked whether they are willing to participate in to the study and to answer one question about their previous neurosurgical treatment. This question is not considered to be burdensome for the patients. Moreover, this study cannot be conducted without the data of these patients and the results are of public importance. Therefore, it is reasonable to proceed with the study without obtaining written informed consent. The results obtained in this study will give important insights in the risk of ASD after different surgical techniques. This might lead to other primary treatment techniques, which might prevent re-operations and hospital admissions for future patients. Before using patients' data, records will be checked for objection to participation in research. All data will be anonymized. A neurosurgeon or resident neurosurgery with a treatment relationship to the patient will contact them by phone to ask for re-operation in a different centre. Patients will not be burdened by this study, as they will only have to reply to one phone call. Patients will not receive a reimbursement for participation.
5. VALORISATION AND PUBLICATION The results of this study will lead to more insights in the reoperation rates for adjacent segment disease in the study population after anterior cervical decompression surgery CDDD. If a relation can be seen between age and Kellgren score and the risk for ASD, a different counselling or treatment choice can be made for this population. If a specific age group seems to have a lower risk on ASD, they might not experience benefit from motion-sparing surgery. Moreover, the investigators might be able to determine a difference in re-operation rates for ASD in different anterior surgical techniques, which can also influence treatment decisions. Results of this study will be submitted to peer-reviewed open access journals. In this publication, data will be anonymized and will also be submitted when they turn out to be negative. None of the involved parties have veto about whether or not data is published.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic single-level or multi-level radiculopathy and/or myelopathy due to CDDD, which corresponds to the afflicted level on radiologic imaging.
* Neurosurgical technique used: anterior cervical discectomy (simple discectomy, ACD), anterior cervical discectomy with fusion (ACDF) with or without plating, corpectomy.
* Minimum age 18 years.
* Adequately documented treatment.
* Follow up data available in electronic patients records for at least one outpatient follow-up visit weeks post-operative

Exclusion Criteria:

* Any other cause than degenerative disc disease for radiculopathy and/or myelopathy such as compression by spinal tumours, trauma, infection or rheumatologic pathologies.
* Objection to participate in scientific research.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients who underwent anterior cervical decompression for radiculopathy and/or myelopathy due to cervical degenerative disc disease in the Zuyderland MC Heerlen or Maastricht UMC+ in the past 10 years. Anterior surgical decompression techniques that will be included are ACD, ACDF, ACDF with plating and corpectomy.
Sampling Method: Non-Probability Sample
Enrollment: 673 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The incidence of re-operation for adjacent segment disease | Available patient records from the primary intervention (10 years in retrospective) until present time will be analysed.
  Assessing whether a patient underwent a re-operation for ASD (yes/no) after the primary intervention for radiculopathy and/or myelopathy due to cervical degenerative disc disease. To determine this, patient records will be analysed.

SECONDARY OUTCOMES:
Radiculopathy: the number of patients with a good outcome and the number of patients with a poor outcome among those who underwent an intervention for radiculopathy. | Available patient records from the primary intervention (10 years in retrospective) until present time will be analysed.
  Measured in patients that underwent primary intervention for cervical radiculopathy due to cervical degenerative disc disease. Assessing whether radiculopathy improved (good outcome) or deteriorated/stabilized (poor outcome), as described by a neurosurgeon or neurosurgical resident in patient records.
Myelopathy: the number of patients with a good outcome and the number of patients with a poor outcome among those who underwent an intervention for myelopathy. | Available patient records from primary intervention (10 years in retrospective) until present time will be analysed.
  Measured in patients that underwent primary intervention for cervical myelopathy due to cervical degenerative disc disease. Assessing whether myelopathy improved/stabilized (good outcome) or deteriorated (poor outcome), as described by a neurosurgeon or neurosurgical resident in patient records.
New symptoms | Available patient records from primary intervention (10 years in retrospective) until present will be analysed.
  Assessing whether patients developed new symptoms (yes/no) after the primary treatment, radiculopathy or myelopathy and the affected level.

OTHER OUTCOMES:
The occurrence of complications related to surgery | Available patient records from primary intervention (10 years in retrospective) until present or death will be analysed.
  Assessing whether complications related to surgery occurred, classified as none/failure of treatment/death.

CONTACTS AND LOCATIONS:
Overall Officials: Henk van Santbrink, MD, PhD, prof, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Zuyderland Medisch Centrum, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nouri A, Tetreault L, Singh A, Karadimas SK, Fehlings MG. Degenerative Cervical Myelopathy: Epidemiology, Genetics, and Pathogenesis. Spine (Phila Pa 1976). 2015 Jun 15;40(12):E675-93. doi: 10.1097/BRS.0000000000000913. PMID 25839387
- [Background] McCartney S, Baskerville R, Blagg S, McCartney D. Cervical radiculopathy and cervical myelopathy: diagnosis and management in primary care. Br J Gen Pract. 2018 Jan;68(666):44-46. doi: 10.3399/bjgp17X694361. No abstract available. PMID 29284641
- [Background] Kuijper B, Tans JT, Beelen A, Nollet F, de Visser M. Cervical collar or physiotherapy versus wait and see policy for recent onset cervical radiculopathy: randomised trial. BMJ. 2009 Oct 7;339:b3883. doi: 10.1136/bmj.b3883. PMID 19812130
- [Background] Saal JS, Saal JA, Yurth EF. Nonoperative management of herniated cervical intervertebral disc with radiculopathy. Spine (Phila Pa 1976). 1996 Aug 15;21(16):1877-83. doi: 10.1097/00007632-199608150-00008. PMID 8875719
- [Background] Fehlings MG, Tetreault LA, Riew KD, Middleton JW, Aarabi B, Arnold PM, Brodke DS, Burns AS, Carette S, Chen R, Chiba K, Dettori JR, Furlan JC, Harrop JS, Holly LT, Kalsi-Ryan S, Kotter M, Kwon BK, Martin AR, Milligan J, Nakashima H, Nagoshi N, Rhee J, Singh A, Skelly AC, Sodhi S, Wilson JR, Yee A, Wang JC. A Clinical Practice Guideline for the Management of Patients With Degenerative Cervical Myelopathy: Recommendations for Patients With Mild, Moderate, and Severe Disease and Nonmyelopathic Patients With Evidence of Cord Compression. Global Spine J. 2017 Sep;7(3 Suppl):70S-83S. doi: 10.1177/2192568217701914. Epub 2017 Sep 5. PMID 29164035
- [Background] Fehlings MG, Kwon BK, Tetreault LA. Guidelines for the Management of Degenerative Cervical Myelopathy and Spinal Cord Injury: An Introduction to a Focus Issue. Global Spine J. 2017 Sep;7(3 Suppl):6S-7S. doi: 10.1177/2192568217701714. Epub 2017 Sep 5. PMID 29164034
- [Background] Dowd GC, Wirth FP. Anterior cervical discectomy: is fusion necessary? J Neurosurg. 1999 Jan;90(1 Suppl):8-12. doi: 10.3171/spi.1999.90.1.0008. PMID 10413119
- [Background] Hilibrand AS, Carlson GD, Palumbo MA, Jones PK, Bohlman HH. Radiculopathy and myelopathy at segments adjacent to the site of a previous anterior cervical arthrodesis. J Bone Joint Surg Am. 1999 Apr;81(4):519-28. doi: 10.2106/00004623-199904000-00009. PMID 10225797
- [Background] Helgeson MD, Bevevino AJ, Hilibrand AS. Update on the evidence for adjacent segment degeneration and disease. Spine J. 2013 Mar;13(3):342-51. doi: 10.1016/j.spinee.2012.12.009. Epub 2013 Feb 15. PMID 23420004
- [Background] Hilibrand AS, Robbins M. Adjacent segment degeneration and adjacent segment disease: the consequences of spinal fusion? Spine J. 2004 Nov-Dec;4(6 Suppl):190S-194S. doi: 10.1016/j.spinee.2004.07.007. PMID 15541666
- [Background] Davis RJ, Kim KD, Hisey MS, Hoffman GA, Bae HW, Gaede SE, Rashbaum RF, Nunley PD, Peterson DL, Stokes JK. Cervical total disc replacement with the Mobi-C cervical artificial disc compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled multicenter clinical trial: clinical article. J Neurosurg Spine. 2013 Nov;19(5):532-45. doi: 10.3171/2013.6.SPINE12527. Epub 2013 Sep 6. PMID 24010901
- [Background] Radcliff K, Lerner J, Yang C, Bernard T, Zigler JE. Seven-year cost-effectiveness of ProDisc-C total disc replacement: results from investigational device exemption and post-approval studies. J Neurosurg Spine. 2016 May;24(5):760-8. doi: 10.3171/2015.10.SPINE15505. Epub 2016 Jan 29. PMID 26824587
- [Background] Radcliff K, Davis RJ, Hisey MS, Nunley PD, Hoffman GA, Jackson RJ, Bae HW, Albert T, Coric D. Long-term Evaluation of Cervical Disc Arthroplasty with the Mobi-C(c) Cervical Disc: A Randomized, Prospective, Multicenter Clinical Trial with Seven-Year Follow-up. Int J Spine Surg. 2017 Nov 28;11(4):31. doi: 10.14444/4031. eCollection 2017. PMID 29372135
- [Background] Joaquim AF, Riew KD. Multilevel cervical arthroplasty: current evidence. A systematic review. Neurosurg Focus. 2017 Feb;42(2):E4. doi: 10.3171/2016.10.FOCUS16354. PMID 28142256